CLINICAL TRIAL: NCT05461170
Title: A Phase 2 Study to Evaluate Efficacy, Safety and Tolerability of VIR-2218 and VIR-3434 in Participants With Chronic Hepatitis D Virus Infection (SOLSTICE)
Brief Title: SOLSTICE: Combination Therapy for the Treatment of Chronic Hepatitis D Infection.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIR-CHDV-V201
Record Dates: First submitted 2022-07-01; First posted 2022-07-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis D, Chronic
Keywords: HDV; Hepatitis D Virus; Hepatitis; Chronic Hepatitis D Virus; Hepatitis Delta Virus
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis; Hepatitis D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Cohort 1a (VIR-2218) (Experimental): Participants will receive multiple doses of VIR-2218 for up to 96 weeks total.
  Interventions: Drug: VIR-2218
- Cohort 1b (VIR-3434) (Experimental): Participants will receive multiple doses of VIR-3434 for up to 96 weeks total.
  Interventions: Drug: VIR-3434
- Cohort 2a (VIR-2218) (Experimental): Participants will receive multiple doses of VIR-2218 for up to 132 weeks, then assign to Cohort 2c.
  Interventions: Drug: VIR-2218
- Cohort 2b1 (VIR-3434) (Experimental): Participants will receive multiple doses of VIR-3434 for up to 132 weeks, then assign to Cohort 2c.
  Interventions: Drug: VIR-3434
- Cohort 2b2 (VIR-3434) (Experimental): Participants will receive multiple doses of VIR-3434 for up to 132 weeks, then assign to Cohort 2c.
  Interventions: Drug: VIR-3434
- Cohort 2c (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for up to 192 weeks.
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 3 (VIR-3434) (Experimental): Participants will receive multiple doses of VIR-3434 for up to 112 weeks, then assign to Cohort 2c.
  Interventions: Drug: VIR-3434
- Cohort 4 (NRTI) (Placebo Comparator): Participants will receive NRTI for 12 weeks, then assign to Cohort 2c or Cohort 3.
  Interventions: Drug: NRTI
- Cohort 5 (VIR-2218) (Experimental): Participants will receive multiple doses of VIR-2218 for 12 weeks, then assign to Cohort 2c.
  Interventions: Drug: VIR-2218

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Other Names: Elebsiran
  Arms: Cohort 1a (VIR-2218); Cohort 2a (VIR-2218); Cohort 2c (VIR-2218 + VIR-3434); Cohort 5 (VIR-2218)
Drug: VIR-3434 — VIR-3434 given by subcutaneous injection
  Other Names: Tobevibart
  Arms: Cohort 1b (VIR-3434); Cohort 2b1 (VIR-3434); Cohort 2b2 (VIR-3434); Cohort 2c (VIR-2218 + VIR-3434); Cohort 3 (VIR-3434)
Drug: NRTI — NRTI given orally.
  Arms: Cohort 4 (NRTI)

SUMMARY:
This is a phase 2 trial in which participants with chronic hepatitis D virus (HDV) infection will receive VIR-2218 and/or VIR-3434 and be assessed for safety, tolerability, and efficacy

DETAILED DESCRIPTION:
Participants may be enrolled into Cohort 1 (1a and 1b) or Cohort 2 (2a, 2b1 or 2b2, 2c), 3, 4, and 5. All participants still receiving VIR-2218 or VIR-3434 monotherapy at the time of implementation of Protocol Amendment 4 will switch to combination therapy at Week 132 (Cohort 2a, 2b1/2b2) or Week 112 (Cohort 3).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 to < 70 years at screening
* Chronic HDV infection for >/= 6 months
* On NRTI therapy for at least 12 weeks prior to day 1
* ALT>ULN and < 5x ULN
* Non-cirrhotic and CPT-A cirrhotic

Exclusion Criteria:

* Any clinically significant chronic or acute medical or psychiatric condition that makes the participant unsuitable for participation.
* History of significant liver disease from non-HBV or non-HDV etiology
* History of allergic reactions, hypersensitivity, or intolerance to study drug, its metabolites, or excipients.
* History of anaphylaxis
* History of immune complex disease
* History of autoimmune disorder
* History or evidence of alcohol or drug abuse
* Prior or concomitant therapy with an immunomodulatory agent, IFN-alpha, cytotoxic or chemotherapeutic agent, or chronic corticosteroids.
* Anti-HBs >10 mIU/mL at screening

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with undetectable HDV RNA (< limit of detection [LOD]) or ≥ 2 log10 decrease in HDV RNA from baseline and alanine aminotransferase (ALT) normalization (ALT < upper limit of normal [ULN]) at Week 24 | Up to 24 Weeks
Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to 118 Weeks

SECONDARY OUTCOMES:
Proportion of participants with undetectable HDV RNA (less than LOD) or greater than/equal to 2 log10 decrease in HDV RNA from baseline and ALT normalization at Week 12, Week 48, Week 72, Week 96, Week 144, and Week 192. | Up to 192 Weeks
Proportion of participants with undetectable HDV RNA (less than LOD) or greater than/equal to 2 log10 decrease in HDV RNA from baseline at Week 12, Week 24, Week 48, Week 72, Week 96, Week 144, and Week 192. | Up to 192 Weeks
Proportion of participants with undetectable HDV RNA (less than LOD) at Week 12, Week 24, Week 48, Week 72, Week 96, Week 144, and Week 192. | Up to 192 Weeks
Proportion of participants with HDV RNA < lower limit of quantitation (LLOQ) at Week 12, Week 24, Week 48, Week 72, Week 96, Week 144, and Week 192. | Up to 192 Weeks
Change from baseline in HDV RNA at Week 12, Week 24, Week 48, Week 72, Week 96, Week 144, and Week 192. | Up to 192 Weeks
Proportion of participants with ALT normalization at Week 12, Week 24, Week 48, Week 72, Week 96, Week 144, and Week 192. | Up to 192 Weeks
Incidence of anti-drug antibodies (ADA) and titers of ADA to VIR-3434 at specified study visits up to Week 192 (for cohorts with VIR3434) | Up to 192 Weeks
Change from baseline in liver fibrosis at Week 48, Week 96, Week 144, and Week 192 | Up to 192 Weeks.
  Liver Fibrosis will be measured by conventional Transient Elastography imaging technique reported in kPa.
Change from baseline in Model for End Stage Liver Disease (MELD) score at Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 144, and Week 192 | Up to 192 Weeks
  MELD score will be calculated using serum bilirubin, serum creatinine, and International Normalized Ratio.
Change from baseline in Child-Pugh-Turcotte (CPT) score at Week 24, Week 48, Week 72, Week 96, Week 144, and Week 192 | Up to 192 Weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Bulgaria (2):
  - Investigative Site, Sofia
  - Investigative Site, Stara Zagora
- France (4):
  - Investigative Site, Clichy
  - Investigative Site, Pessac
  - Investigative Site, Rennes
  - Investigative Site, Toulouse
- Germany (3):
  - Investigative Site, Frankfurt
  - Investigative Site, Hanover
  - Investigative Site, Tübingen
- Italy (2):
  - Investigative Site, Milan
  - Investigative Site, Pisa
- Investigative Site, Chisinau, Moldova
- Investigative Site, Rotterdam, Netherlands
- Investigative Site, Auckland, New Zealand
- Investigative Site, Bucharest, Romania
- United Kingdom (3):
  - Investigative Site, Birmingham
  - Investigative Site, London
  - Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asselah T, Chattergoon MA, Jucov A, Streinu-Cercel A, Lampertico P, Wedemeyer H, Kennedy PT, Gane EJ, Bullard BL, Chow S, Santos D, Camus G, Lu Y, Pilowa C, Hwang C, Correll T, Agarwal K; SOLSTICE Trial Investigators. A Phase 2 Trial of Tobevibart plus Elebsiran in Hepatitis D. N Engl J Med. 2026 Jan 22;394(4):343-353. doi: 10.1056/NEJMoa2508827. Epub 2025 Nov 9. PMID 41211943